CLINICAL TRIAL: NCT02646306
Title: A New Neurocognitive Interpretation of the Shoulder Position Sense During Reaching
Brief Title: A New Shoulder Proprioceptive Rehabilitative Tool (SRPT) for the Evaluation of the Role of the Shoulder During Reaching
Acronym: SRPT-Iphase
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Director, University of Roma La Sapienza
Other Study IDs: 3826/2015
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-01

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder; proprioception; movement; reaching
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Shoulder Impingement Syndrome: Execution of two tests in succession with the use of the shoulder proprioceptive rehabilitation tool (SRPT), each oriented to indicate a specific discriminative and integrative mode in the movement of the scapulothoracic. Will be required to each subject to perform recognition tasks that include both retraction movements of the hand, starting from a start position, and approaching movements of the hand, starting from an end position. First test: ability to integrate visual and proprioceptive informations. Second test: discriminative proprioceptive capacity of the subject, thus excluding the contribution of the view.
  Interventions: Other: shoulder proprioceptive rehabilitation tool
- Healthy Subjects: Execution of two tests in succession with the use of the shoulder proprioceptive rehabilitation tool (SRPT), each oriented to indicate a specific discriminative and integrative mode in the movement of the scapulothoracic. Will be required to each subject to perform recognition tasks that include both retraction movements of the hand, starting from a start position, and approaching movements of the hand, starting from an end position. First test: ability to integrate visual and proprioceptive informations. Second test: discriminative proprioceptive capacity of the subject, thus excluding the contribution of the view.
  Interventions: Other: shoulder proprioceptive rehabilitation tool

INTERVENTIONS:
Other: shoulder proprioceptive rehabilitation tool — Using of this tool to measure which is the average error in reaching back in both healthy subjects and subjects with shoulder impingement syndrome starting from the assumption that the shoulder, through the articulation scapulothoracic, helps to determine direction and distance during the "reaching" of an object.
  Other Names: SRPT

SUMMARY:
The aim of the study focused on the creation of a rehabilitative measuring device (SRPT-shoulder proprioceptive rehabilitation tool) and the development of the examination methodology for assessing the proprioception of the glenohumeral joint respect to scapula abduction, within the movement of antepulsion on the sagittal plane both in healthy subjects and in patients with shoulder impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Diagnosis of subacromial right impingement syndrome performed by the orthopedic specialist (nuclear magnetic resonance and/or ultrasound examination)
* Neer stages 1, 2 and 3
* Presence of pain 3 <VAS<8 at baseline
* Age between 55 and 65 years.

Exclusion Criteria:

* Diabetes mellitus
* Inflammatory systemic diseases
* CNS and/or PNS diseases
* Systemic infectious diseases
* Neoplastic diseases
* Assumption of antidepressants and/or anxiolytics and/or other medications that can affect attention and sensory
* Visual problems not properly compensated
* Previous surgery to the shoulder

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects affected by shoulder impingement syndrome and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Visual Analogue Scale (VAS) at baseline | baseline
  It is an instrument that enables patients to express their pain intensity as a numerical value. Patients were asked to mark the point that corresponded to their perceived pain intensity on a 10-cm line, with 0 indicating the absence of pain and 10 reflecting the most severe pain

SECONDARY OUTCOMES:
Evaluation of the short form of the Disabilities of the Arm, Shoulder and Hand questionnaire (Quick-DASH) at baseline | baseline
  The short form (11 item) of the Disabilities of the Arm, Shoulder and Hand questionnaire (Quick-DASH) measures physical ability and symptoms of the upper extremity and explores the impact of functional impairment and pain on daily-living tasks, as well as on social and recreational activities, work and sleep. The score ranges from 0 to 100 points, with 0 reflect- ing no disability and 100 corresponding to the most severe disability
Evaluation of the Constant-Murley shoulder outcome score at baseline | baseline
  It is based on subjective (sleep, work, and recreational activities) and objective (ROM and strength) components, adjusted for age and sex, according to normative values reported by Yian et al. The score ranges from 0 (worst result) to 100 (best result).

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Principal Investigator — Umberto I Hospital, University "Sapienza" of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy